CLINICAL TRIAL: NCT02538094
Title: Transcranial Direct Current Stimulation and Cognition in Adults With Multiple Sclerosis or Encephalitis
Brief Title: tDCS and Cognition in Adults With Multiple Sclerosis or Encephalitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00033581
Record Dates: First submitted 2015-03-25; First posted 2015-09-02 (Estimated); Results first posted 2020-04-06 (Actual); Last update posted 2020-04-06 (Actual); Status verified 2020-04

CONDITIONS: Multiple Sclerosis; Encephalitis
Keywords: Cognitive Enhancement; tDCS; stimulation; MS; Multiple Sclerosis; Encephalitis
MeSH Terms: conditions — Multiple Sclerosis; Encephalitis | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sham Stimulation First (Sham Comparator): Transcranial direct current stimulation (tDCS) that is ramped up and ramped down providing the sensation of tDCS without delivering the full amount of tDCS first and then Anodal Stimulation second.
  Interventions: Device: Sham Transcranial direct current stimulation; Device: Anodal Transcranial direct current stimulation
- Anodal Stimulation First (Experimental): Transcranial direct current stimulation using Anodal stimulation first over the area of interest and then Sham Stimulation second.
  Interventions: Device: Sham Transcranial direct current stimulation; Device: Anodal Transcranial direct current stimulation

INTERVENTIONS:
Device: Sham Transcranial direct current stimulation — Delivery of sham stimulation for 30 minutes using Neuro-Conn Direct Current (DC) Stimulator Plus.
  Other Names: tDCS
Device: Anodal Transcranial direct current stimulation — Delivery of transcranial direct current stimulation for 30 minutes.
  Other Names: tDCS

SUMMARY:
This research is being done to determine whether transcranial direct current stimulation (tDCS) can improve certain mental abilities in individuals with multiple sclerosis (MS) or encephalitis. Participants will be asked to come in daily for two full weeks during which time participants will undergo cognitive testing and Magnetic Resonance Imaging (MRI) brain scans. In this research, a very weak electrical current is administered to the surface of the scalp while participants complete cognitive tasks. The investigators' aim is to find out whether tDCS will improve task performance in adults with multiple sclerosis or encephalitis.

DETAILED DESCRIPTION:
Participants enrolled into this study may be asked to do the following:

* Come to the investigators' testing office at the Johns Hopkins Hospital where the tDCS equipment is located for 10 study visits.
* Grant permission for the researchers to view medical records associated with the participant's diagnosis of multiple sclerosis or encephalitis (if applicable) and general state of health.
* Complete a questionnaire and provide a health history in order to verify eligibility to participate and be able to safely undergo the experimental procedures.
* Complete several computerized, written, and/or aural tasks (i.e., saying words out loud) that assess different cognitive functions such as attention, memory, language, or processing speed.
* Wear electrodes that will be placed on the scalp with a large rubberized band. These electrodes will administer very weak electrical current (tDCS) for 30 minutes.
* Participate in several study conditions. The exact conditions and the order will be randomized. That is, the conditions and order will vary by chance (like the flip of a coin). Under some conditions, the participant might receive active stimulation (tDCS) and under other conditions, the participant might receive placebo (or sham) stimulation. Placebo stimulation is similar to active tDCS but lasts only a few seconds. However, all groups will wear the electrodes for the same length of time to prevent the participant from knowing whether participants are receiving active tDCS or sham stimulation. The study doctor and research staff will know which group the participant is in.
* Permission to audio and/or video-tape test sessions for later scoring and observation. These tapes will not be viewed by anyone not affiliated with the study without the participant's consent.
* Have structural, resting-state and functional Magnetic Resonance Imaging scans as a part of the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of multiple sclerosis or encephalitis
* Over the age of 18

Exclusion Criteria:

* A diagnosis of schizophrenia bipolar disorder
* Beck Depression Inventory-II scores over 20
* Mini Mental Exam below 24
* Any uncontrolled seizure disorder
* Any implanted metal device or hearing aids
* Use of medication shown to interact with tDCS effectiveness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2014-09; Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tracy Vannorsdall, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins East Baltimore Campus; Medical Psychiatry department, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Sham tDCS First: Participants received sham tDCS first and then active anodal tDCS after washout.
- Active Anodal tDCS First: Participants received active anodal tDCS first and then sham tDCS after washout.
Period: Intervention 1 (5 Days Per Participant)
Arm/Group | Sham tDCS First | Active Anodal tDCS First
Started | 2 | 5
Completed | 2 | 4
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Washout (4 Weeks)
Arm/Group | Sham tDCS First | Active Anodal tDCS First
Started | 2 | 4
Completed | 2 | 3
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Intervention 2 (5 Days Per Participant)
Arm/Group | Sham tDCS First | Active Anodal tDCS First
Started | 2 | 3
Completed | 2 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: Transcranial direct current stimulation using Anodal stimulation over the area of interest or sham stimulation using Neuro-Conn Direct Current (DC) Stimulator Plus.
Arm/Group | All Participants
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.29 (11.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7
Paced Auditory Serial Addition Test [Mean (Standard Deviation); unit: score on a scale] — The Paced Auditory Serial Addition Test (PASAT) is a measure of cognitive function that assesses auditory information processing speed and flexibility, as well as calculation ability. PASAT scores range from 0 to 120 with higher scores reflecting better performance.
  score on a scale | 76.29 (25.21)
Multidimensional Fatigue Symptom Inventory 30-item short form score [Mean (Standard Deviation); unit: score on a scale] — The Multidimensional Fatigue Symptom Inventory 30-item short form (MFSI-SF) is an instrument for assessing fatigue. MFSI-SF scores range from 0 to 84, with higher values reflecting greater fatigue.
  score on a scale | 55.43 (23.06)

OUTCOME MEASURES:

1. Primary Outcome: Change in Cognition as Assessed by Change in Paced Auditory Serial Addition Test Scores
Description: Change in performance on an individual cognitive test measure raw score from the Minimal Assessment of Cognitive Function in Multiple Sclerosis (MACFIMS) battery tests (i.e. Paced Auditory Serial Addition Test scores). Change scores range from -120 to + 120. Positive change scores reflect improvement at the end of the intervention relative to baseline. Negative change scores reflect decline at the end of the intervention relative to baseline.
Time Frame: Assessed at beginning and end of a 5-day treatment week
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Sham tDCS: Sham transcranial direct current stimulation (tDCS) is ramped up and ramped down providing the sensation of tDCS without delivering the full amount of tDCS. Delivery of sham stimulation using Neuro-Conn Direct Current (DC) Stimulator Plus.
- Active Anodal tDCS: Active transcranial direct current stimulation using anodal stimulation over the area of interest. Delivery of transcranial direct current stimulation for 30 minutes.
Arm/Group | Sham tDCS | Active Anodal tDCS
Number analyzed (Participants) | 5 | 6
score on a scale | -1.20 (6.26) | -0.33 (9.42)

2. Secondary Outcome: Change in Fatigue as Assessed by Multidimensional Fatigue Symptom Inventory 30-item Short Form (MFSI-SF) Total Scores
Description: Fatigue was measured via changes in self-reported fatigue on the Multidimensional Fatigue Symptom Inventory 30-item short form (MFSI-SF) total score over the course of active and sham tDCS. Change scores range from -84 to + 84. Positive change values reflect increased symptom burden at the end of the intervention relative to baseline. Negative change scores reflect reduced symptom burden at the end of the intervention relative to baseline.
Time Frame: Assessed at beginning and end of a 5-day treatment week
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sham tDCS | Active Anodal tDCS
Number analyzed (Participants) | 5 | 6
score on a scale | -7.40 (8.08) | -15.0 (18.23)

ADVERSE EVENTS:
Time Frame: Up to 6 weeks
Arm/Group | Sham tDCS | Active Anodal tDCS
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/7
Other Adverse Events (participants affected / at risk) | 0/6 | 0/7

LIMITATIONS AND CAVEATS:
Recruitment was not sufficient to permit planned statistical analyses.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-02-28): https://cdn.clinicaltrials.gov/large-docs/94/NCT02538094/Prot_SAP_000.pdf
  • Informed Consent Form (2016-11-11): https://cdn.clinicaltrials.gov/large-docs/94/NCT02538094/ICF_001.pdf